CLINICAL TRIAL: NCT04639063
Title: Clinico-pathological Assessment of Surgically Removed Abdominal Wall Endometriomas
Brief Title: Assessment of Surgically Removed Abdominal Wall Endometriomas
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdulkarim Hasan, Pathologist and Laboratory Director, Al-Azhar University
Other Study IDs: PMS20-11-01
Record Dates: First submitted 2020-11-17; First posted 2020-11-20 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Endometriosis Outside Pelvis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cesarean sectioned: All females who treated in our hospital by Cesarean section operation during two-years-period
- Complicated with Abdominal wall endometriosis: All the surgically excised endometrioma cases during the same time period
  Interventions: Other: Microscopic examination using H&E stained slides

INTERVENTIONS:
Other: Microscopic examination using H&E stained slides — Reexamination of the stained slides of the patients from the hospital archive and adding a CD10 stain when required
  Other Names: CD10 immunohistochemistry
  Groups: Complicated with Abdominal wall endometriosis

SUMMARY:
A retrospective review of all patients who underwent surgery for an anterior abdominal wall mass which confirmed by pathology examination as an endometrioma will be completely performed. The clinical data will be recorded and pathology report diagnosis will be correlated with the clinical data to assess the possible causes of endometrioma in the women treated in our tertiary hospital and the efficacy of the surgical excision.

DETAILED DESCRIPTION:
Our hospital is a tertiary center for performing Cesarean sections, external endometriosis (Endometrioma) is a challenging complication for this operation, many treatment choices are available and the most common is the surgical excision, however recurrence could be seen after the surgical operation. We assess all patients who underwent surgical excision for abdominal wall endometriomas in our hospital by retrieving the medical files and pathology reports to study the possible age group,causes and duration of endometriomas. Also the rate of enodmetriomas among the previously experienced females with cesarean section operations. Pathological diagnosis tools will be also assessed.

Ethical approval was obtained from the local committee. Results will be statistically assessed using SPSS programm.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Surgically removed abdominal wall endometrioma

Exclusion Criteria:

* Male (very very rare to occur)
* medically treated enodmetrioma
* Outside treated patients

Ages: 15 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female patients treated in our hospital and pathologically examined in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Positive for endometrioma | 1 day
  Presence of endometrial glands and stroma along with hemosidren pigment under microscopic examination, confirms the diagnosis and the case will be calculated and the related clinical data

CONTACTS AND LOCATIONS:
Overall Officials: Abdulkarim Hasan, MD, Principal Investigator — Al-Azhar University
Locations (1):
- Abdulkarim Hasan, Cairo, Egypt